CLINICAL TRIAL: NCT04688593
Title: Clinical and Functional Outcome of the MobileLink Acetabular Cup System in the Short-, Mid-, and Longterm Follow-up
Status: Recruiting | Type: Observational
Sponsor: Waldemar Link GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: HP15
Record Dates: First submitted 2020-12-16; First posted 2020-12-30 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis, Hip; Hip Osteoarthritis; Prosthesis Survival; Prosthesis Failure
Keywords: MobileLink
MeSH Terms: conditions — Osteoarthritis, Hip; Prosthesis Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: MobileLink — Patients who receive a MobileLink hip prosthesis system will be followed-up for 10 years.

SUMMARY:
The implantation of artificial hip joints is one of the most frequently performed surgeries. Normally, patients are very satisfied with the results.

The MobileLink hip prosthesis system is a CE marked medical device. This means the the safety and performance of the prosthesis ist approved. Aim of the study is to collect clinical data about the outcome of the MobileLink hip prosthesis system under routine condition and to determine the satisfaction of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Implantation of a MobileLink acetabular cup system and a femoral stem manufactured by Waldemar Link
* Age ≥ 18 years
* Fully signed patient informed cons

Exclusion Criteria:

* Revisions
* Body Mass Index (BMI) ≥ 40 kg/m²
* Patient who is foreseeable not able to understand the study and the study-related circumstances
* Patients who is foreseeable non-compliant to the treatment and the follow-ups
* Pregnant or breast-feeding women
* Prisoner

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2036-01 (Estimated); Study Completion 2036-01 (Estimated)

PRIMARY OUTCOMES:
Survival rate of the complete MobileLink hip prosthesis system with revision for any reason as the endpoint, | 10-years
  calculated with Kaplan-Meier method.

SECONDARY OUTCOMES:
Revision rates of the complete MobileLink acetabular cup system with revision for any reason except peri-prosthetic infections as the endpoint | 3 months, 1 year, 3, 5, 7 and 10 years
Revision rates of the MobileLink acetabular cup system shell(s) with revision for any reason as the endpoint | 3 months, 1 year, 3, 5, 7 and 10 years
Revision rates of the MobileLink acetabular cup system inserts (Ceramic, XLINKed, E-Dur) with revision for any reason as the endpoint | 3 months, 1 year, 3, 5, 7 and 10 years
Revision rates of the combined LINK hip stem(s) with revision for any reason as the endpoint | 3 months, 1 year, 3, 5, 7 and 10 years
Change of baseline hip functionality | pre-operatively and at the 3 months, 1 year, 3, 5, 7 and 10 year follow-up
  measured by the Harris Hip Score (HHS) (maximum 100 points, minimum 0 points, a higher score indicates a better outcome)
Change of baseline hip functionality | pre-operatively and at the 3 months, 1 year, 3, 5, 7 and 10 year follow-up
  measured by the Hip disability and osteoarthritis outcome score (HOOS), (maximum 100 points, minimum 0 points, a higher score indicates a better outcome)
Rate of complications and re-operations of the hip joint | 3 months, 1 year, 3, 5, 7 and 10 year follow-up
Rate of failed osteointegrated cups | 3 months, 1 year, 3, 5, 7 and 10 year follow-up
  radiological assessment
Rate of failed osteointegrated stems | 3 months, 1 year, 3, 5, 7 and 10 year follow-up
  radiological assessment
Change of postoperative cup position | 3 months, 1 year, 3, 5, 7 and 10 year follow-up
  radiological assessment
Change of postoperative stem position | 3 months, 1 year, 3, 5, 7 and 10 year follow-up
  radiological assessment
Occurence of heterotopic ossifications | 3 months, 1 year, 3, 5, 7 and 10 year follow-up
  radiological assessment, classified according to Brooker
Type and rate of complications with the used instruments related to usability and sterilization | intraoperatively
Survival rate of the complete MobileLink hip prosthesis system with revision for any reason as the endpoint | 3 month
  calculated with Kaplan-Meier method.
Survival rate of the complete MobileLink hip prosthesis system with revision for any reason as the endpoint | 1 year
  calculated with Kaplan-Meier method.
Survival rate of the complete MobileLink hip prosthesis system with revision for any reason as the endpoint | 3 year
  calculated with Kaplan-Meier method.
Survival rate of the complete MobileLink hip prosthesis system with revision for any reason as the endpoint | 5 year
  calculated with Kaplan-Meier method.
Survival rate of the complete MobileLink hip prosthesis system with revision for any reason as the endpoint | 7 year
  calculated with Kaplan-Meier method.
Survival rate of the complete MobileLink hip prosthesis system with revision for any reason as the endpoint | 10 year
  calculated with Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Locations (2):
- Lubinus Stiftung, Kiel, Germany
- NHS FIFE Victoria Hospital, Kirkcaldy, United Kingdom